CLINICAL TRIAL: NCT04286815
Title: Gene Therapy for X Linked Severe Combined Immunodeficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, mingfeng hu, Resident physician, Children's Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHCMU gene therapy
Record Dates: First submitted 2020-02-23; First posted 2020-02-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Gene Therapy
Keywords: Gene Therapy; X Linked Severe Combined Immunodeficiency; Lentiviral Vector
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): a lentiviral vector to transfer IL2RG complementary DNA to bone marrow stem cells in ten children with genetic diagnosed X-SCID（severe combined immune deficiency）.
  Interventions: Device: Lentiviral Vector Gene Therapy

INTERVENTIONS:
Device: Lentiviral Vector Gene Therapy — Lentiviral vector to transfer IL2RG complementary DNA to patients'bone marrow stem cells

SUMMARY:
A safety and efficacy clinical study of a lentiviral vector to transfer IL2RG complementary DNA to bone marrow stem cells in ten children with genetic diagnosed X-SCID（severe combined immune deficiency ）.The ten children will be followed for 3-5 years and be evaluated by clinical characteristics, vector marking (vector copy number per cell) in blood and bone marrow cells, immune reconstitution vector insertion-site patterns and so on.

ELIGIBILITY:
Inclusion Criteria:

1. X-SCID patients diagnosed by IL2RG single gene mutation
2. No HLA（human leukocyte antigen） matching donor
3. Hematopoietic stem cell transplantation failed and the time from transplantation was more than 18 months
4. Severe and persistent refractory infections
5. Life expectancy of > : 4 months
6. HIV PCR in peripheral blood was negative
7. the children and their families signed informed consent and were willing to enter the clinical trial and complete follow-up

Exclusion Criteria:

1. The patient has diagnosed with hematological malignant diseases
2. Received chemotherapy within 3 months
3. HIV infection or HBV（hepatitis B virus） infection
4. The patient or his first-degree relative has developed a malignant tumor within the age of 18 or has been diagnosed with malignant tumor prone genes
5. Although the patient with X-SCID was diagnosed as IL2RG single gene mutation , the clinical phenotype was not severe, so they could continue to wait for the donor search;
6. Patients whose family members have no intention to continue the follow-up treatment in any link

Max Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
1-year survival rate 1-year survival rate | one year after gene therapy of last recruited patient
  1-year survival rate of 10 recruited patients
3-year survival rate | three years after gene therapy of last recruited patient
  3-year survival rate of 10 recruited patients
5-year survival rate | five years after gene therapy of last recruited patient
  5-year survival rate of 10 recruited patients

SECONDARY OUTCOMES:
Growth velocity after gene therapy,weight in kilograms, height in meters | through study completion, an average of 2 year
  Body weight and height of patients will be assessed prior to (month 0) and post gene therapy,weight in kilograms, height in meters
Vector marking (vector copy number per cell) in blood and bone marrow cells | through study completion, an average of 1 year
  vector marking in T cells, B cells, NK cells, myeloid cells, and bone marrow progenitors.
Absolute numbers of peripheral-blood immune-cell subsets | through study completion, an average of 1 year
  Absolute numbers of peripheral-blood immune-cell subsets，as determined by means of standard flow cytometry
Quantity of DNA T-cell-receptor excision circles (TRECs) in peripheral-blood mononuclear cells | through study completion, an average of 1 year
  Quantity of DNA T-cell-receptor excision circles (TRECs) in peripheral-blood ，as determined by means of quantitative polymerase chain reaction (PCR)
Serum immunoglobulins levels | through study completion, an average of 2 year
  Serum immunoglobulins levels will be reported IgM（immunoglobulin M） in mg/dL Serum immunoglobulins levels will be reported IgM in mg/dL
Number of patients without intravenous immune globulin supplementation | through study completion, an average of 2 year
  Number of patients without intravenous immune globulin supplementation after gene therapy
Number of patients who has a response to vaccines | through study completion, an average of 2 year
  Number of patients who has a response to vaccines after gene therapy
Number of patients who recovers from previous infection（virus and bacteria） | through study completion, an average of 2 year
  Number of patients who recovers from previous infection（virus and bacteria）after gene therapy

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Zhao, PHD, Study Director — Assistant President of Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mamcarz E, Zhou S, Lockey T, Abdelsamed H, Cross SJ, Kang G, Ma Z, Condori J, Dowdy J, Triplett B, Li C, Maron G, Aldave Becerra JC, Church JA, Dokmeci E, Love JT, da Matta Ain AC, van der Watt H, Tang X, Janssen W, Ryu BY, De Ravin SS, Weiss MJ, Youngblood B, Long-Boyle JR, Gottschalk S, Meagher MM, Malech HL, Puck JM, Cowan MJ, Sorrentino BP. Lentiviral Gene Therapy Combined with Low-Dose Busulfan in Infants with SCID-X1. N Engl J Med. 2019 Apr 18;380(16):1525-1534. doi: 10.1056/NEJMoa1815408. PMID 30995372
- [Background] Hacein-Bey-Abina S, Hauer J, Lim A, Picard C, Wang GP, Berry CC, Martinache C, Rieux-Laucat F, Latour S, Belohradsky BH, Leiva L, Sorensen R, Debre M, Casanova JL, Blanche S, Durandy A, Bushman FD, Fischer A, Cavazzana-Calvo M. Efficacy of gene therapy for X-linked severe combined immunodeficiency. N Engl J Med. 2010 Jul 22;363(4):355-64. doi: 10.1056/NEJMoa1000164. PMID 20660403
- [Background] De Ravin SS, Wu X, Moir S, Anaya-O'Brien S, Kwatemaa N, Littel P, Theobald N, Choi U, Su L, Marquesen M, Hilligoss D, Lee J, Buckner CM, Zarember KA, O'Connor G, McVicar D, Kuhns D, Throm RE, Zhou S, Notarangelo LD, Hanson IC, Cowan MJ, Kang E, Hadigan C, Meagher M, Gray JT, Sorrentino BP, Malech HL, Kardava L. Lentiviral hematopoietic stem cell gene therapy for X-linked severe combined immunodeficiency. Sci Transl Med. 2016 Apr 20;8(335):335ra57. doi: 10.1126/scitranslmed.aad8856. PMID 27099176